CLINICAL TRIAL: NCT03207035
Title: Effect of Local Anaesthetic Dilution on the Characteristics of Ultrasound Guided Axillary Brachial Plexus Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cork University Hospital (Other)
Responsible Party: Principal Investigator, Dr Anil Ranganath, Dr (Fellow in Regional Anaesthesia), Cork University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ECM 4 (mm)
Record Dates: First submitted 2017-05-07; First posted 2017-07-02 (Actual); Results first posted 2021-10-18 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Brachial Plexus Blockade

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 20 ml of lidocaine 2% with epinephrine (Active Comparator): Patients will receive axillary brachial plexus block with 20 ml of lidocaine 2% with epinephrine.
  Interventions: Procedure: Axillary brachial plexus block
- 40 ml 0f lidocaine 1% with epinephrine (Experimental): Patients will receive axillary brachial plexus block with 20 ml of lidocaine 1% with epinephrine diluted with 20 ml of nacl 0.9% ( total 40 ml)
  Interventions: Procedure: Axillary brachial plexus block

INTERVENTIONS:
Procedure: Axillary brachial plexus block — Ultrasound guided axillary brachial plexus block with local anaesthetic lidocaine with epinephrine

SUMMARY:
We propose to compare the effects of local anaesthetic dilution on the characteristics of the ultrasound guided axillary brachial plexus block.

Administration of 40ml lidocaine 1% with epinephrine will shorten the onset time of ultrasound guided axillary brachial plexus block when compared to 20 mL lidocaine 2% with epinephrine for elective upper limb surgical procedures.

DETAILED DESCRIPTION:
To compare the effects of local anaesthetic 20 mL lidocaine 1% with epinephrine vs 40 mL lidocaine 1% with epinephrine on the onset of sensory and motor block following ultrasound guided axillary brachial plexus block.

Methods:

It is a prospective, randomized, observer blinded study. With institutional ethical approval and having obtained written informed consent from each, 20 patients will be studied.

Randomisation and blinding:

Using a computer generated and sealed envelope technique, 20 patients will be randomly allocated in to one of two groups.

Group 1: patients will receive 20 ml of lidocaine 2% with epinephrine. Group 2: patients will receive 40 ml of lidocaine 1% with epinephrine.

Sample size and statistical analysis:

In the absence of data from previous study using 20 ml of lidocaine with epinephrine for ultrasound guided axillary brachial plexus block. Sample size was calculated based on from our pilot study of 12 patients. We found mean onset of block of 11.25 (SD, 2.3) mins. The minimum sample size required to have an 80% probability of detecting a 30% decrease in onset time (level of significance 0.05) will be 7 patients per group using an unpaired student's t test. Recruited 10 per group

Anaesthetic procedure:

Having established intravenous access, standard anaesthetic monitoring will be applied. Premedication with midazolam will be administered as clinically indicated (to a maximum of 3 mg). The operative arm will be abducted and externally rotated with elbow flexed at 90 degrees. Under strict aseptic condition, ultrasound guided axillary brachial plexus block will be performed. Having identified musculocutaneous, median, radial and ulnar nerves, a 50mm 24-gauge stimuplex short bevel insulated needle will be used with in-plane approach to block each nerve with either 5 (Group 1) or 10 ml (Group 2). All blocks will be performed by operator experienced in the ultrasound peripheral nerve blocks.

Block assessment:

When the block procedure has been completed, a blinded observer will assess the onset of sensory and motor block in the innervation of each nerve every 2.5 mins, until surgical anaesthesia is achieved or 30 mins have elapsed (Table 1). Surgical anaesthesia will be defined as a motor score ≤2, with absent sensation to cold and pinprick. Each nerve distribution will be individually assessed. Onset time will be measured from conclusion of the block (t=0) to attainment of surgical anaesthesia. Block will be deemed failure if surgical anaesthesia has not been achieved at 30 mins in one or more of the four nerve distribution. In case of failure, an additional rescue block or conversion to general anaesthesia will be performed. DATA from these patients will be analysed separately.

Intraoperative period:

All patients will receive 1 g of paracetamol and diclofenac 75 mg iv during surgery. In case of patients discomfort sedation and rescue analgesia in the form of fentanyl 25 micrograms aliquots IV will be administered to a maximum of 100 micrograms.

Postoperative period:

Upon arrival to recovery room, sensory and motor function will be assessed every 15 mins by a blinded observer.15 Assessment will be performed for each nerve separately. Block regression is defined as a return of sensation to cold and pinprick with motor power score ≥3 in any nerve region. Time to first request for postoperative analgesia and total opioid consumption for 24 hrs will be noted. Postoperative analgesia will be prescribed as paracetamol 1 g 6 hourly and diclofenac sodium 75 mg 12 hourly. Oxycodone 5-10 mg orally 4-6 hourly will be administered as rescue analgesia.

Primary Outcome: onset of block.

Secondary Outcomes: Duration of sensory and motor block and block performance data (Imaging time, Needling time, Performance time, No of needle pass, Vascular puncture and parasthesia)

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3
* Patients aged >18 years undergoing elective upper limb (forearm or hand) surgical procedures.

Exclusion Criteria:

* Contraindications to regional anaesthesia
* Hypersensitivity to amide local anaesthetics.
* Chronic pain
* Language barrier
* Neuromuscular disorders or peripheral neuropathy
* Body mass index > 35
* History of hepatic and renal insufficiency
* Pregnancy
* Cognitive or psychiatric disorder
* Cardiac conduction abnormality.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-10-15 (Actual); Primary Completion 2016-03-14 (Actual); Study Completion 2016-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anil Ranganath, FCAI, Principal Investigator — Cork University Hospital

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment
  Assessed for eligibility: n=45 Excluded : n= 25
  * Not meeting inclusion criteria: n = 5
  * Declined to participate: n = 20
  Randomized: n= 20
Period: Overall Study
Arm/Group | 20 ml of Lidocaine 2% With Epinephrine | 40 ml 0f Lidocaine 1% With Epinephrine
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 20 ml of Lidocaine 2% With Epinephrine | 40 ml 0f Lidocaine 1% With Epinephrine | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (18.2) | 48 (15.7) | 47.4 (16.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 7 | 8 | 15
Region of Enrollment [Count of Participants; unit: Participants]
  Ireland | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Onset of Axillary Block
Description: Time taken for onset of sensory and motor axillary brachial plexus block
Time Frame: 1 day
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | 20 ml of Lidocaine 2% With Epinephrine | 40 ml 0f Lidocaine 1% With Epinephrine
Number analyzed (Participants) | 10 | 10
minutes | 8.75 [7.5 to 10] | 6.25 [5 to 7.5]
Statistical Analysis 1: Comparison: 20 ml of Lidocaine 2% With Epinephrine vs 40 ml 0f Lidocaine 1% With Epinephrine; Test type: Other; p = 0.03, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Duration of Sensory and Motor Block
Description: Total duration of sensory and motor block of ultrasound guided axillary brachial plexus block
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 20 ml of Lidocaine 2% With Epinephrine | 40 ml 0f Lidocaine 1% With Epinephrine
Number analyzed (Participants) | 10 | 10
minutes | 165.1 (5.9) | 150.9 (17.2)
Statistical Analysis 1: Comparison: 20 ml of Lidocaine 2% With Epinephrine vs 40 ml 0f Lidocaine 1% With Epinephrine; Test type: Other; p = 0.02, t-test, 2 sided

3. Secondary Outcome: Block Performance Data- Imaging Time
Description: Time taken to obtain appropriate ultrasound image to perform the axillary plexus block
Time Frame: 1 Hour
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 20 ml of Lidocaine 2% With Epinephrine | 40 ml 0f Lidocaine 1% With Epinephrine
Number analyzed (Participants) | 10 | 10
minutes | 2.5 (0.5) | 2.4 (0.6)
Statistical Analysis 1: Comparison: 20 ml of Lidocaine 2% With Epinephrine vs 40 ml 0f Lidocaine 1% With Epinephrine; Test type: Other; p = 0.70, t-test, 2 sided

4. Secondary Outcome: Needling Time
Description: Time taken to perform the block in minutes
Time Frame: 1Hour
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 20 ml of Lidocaine 2% With Epinephrine | 40 ml 0f Lidocaine 1% With Epinephrine
Number analyzed (Participants) | 10 | 10
minutes | 8.5 (1.2) | 6.7 (0.9)
Statistical Analysis 1: Comparison: 20 ml of Lidocaine 2% With Epinephrine vs 40 ml 0f Lidocaine 1% With Epinephrine; Test type: Other; p = 0.002, t-test, 2 sided

5. Secondary Outcome: Performance Time
Description: Sum of imaging and performance time
Time Frame: 1 Hour
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 20 ml of Lidocaine 2% With Epinephrine | 40 ml 0f Lidocaine 1% With Epinephrine
Number analyzed (Participants) | 10 | 10
minutes | 10.9 (1.3) | 9.1 (0.5)
Statistical Analysis 1: Comparison: 20 ml of Lidocaine 2% With Epinephrine vs 40 ml 0f Lidocaine 1% With Epinephrine; Test type: Other; p = 0.001, t-test, 2 sided

6. Secondary Outcome: No of Needle Pass
Description: Number of needle passes while performing the axillary block
Time Frame: 1 Hour
Measure: Mean (Standard Deviation); unit: Needle passes
Arm/Group | 20 ml of Lidocaine 2% With Epinephrine | 40 ml 0f Lidocaine 1% With Epinephrine
Number analyzed (Participants) | 10 | 10
Needle passes | 10.5 (2.3) | 9.1 (0.5)
Statistical Analysis 1: Comparison: 20 ml of Lidocaine 2% With Epinephrine vs 40 ml 0f Lidocaine 1% With Epinephrine; Test type: Other; p = 0.001, t-test, 2 sided

7. Secondary Outcome: Vascular Puncture
Description: Incidence of vascular puncture during the performance of block.
Time Frame: 1 Hour
Measure: Number; unit: participants
Arm/Group | 20 ml of Lidocaine 2% With Epinephrine | 40 ml 0f Lidocaine 1% With Epinephrine
Number analyzed (Participants) | 10 | 10
participants | 2 | 1
Statistical Analysis 1: Comparison: 20 ml of Lidocaine 2% With Epinephrine vs 40 ml 0f Lidocaine 1% With Epinephrine; Test type: Other; p = 0.53, Chi-squared

8. Secondary Outcome: Parasthesia
Description: Incidence of parasthesia during the performance of axillary block
Time Frame: 1 Hour
Measure: Number; unit: Parasthesia events
Arm/Group | 20 ml of Lidocaine 2% With Epinephrine | 40 ml 0f Lidocaine 1% With Epinephrine
Number analyzed (Participants) | 10 | 10
Parasthesia events | 4 | 2
Statistical Analysis 1: Comparison: 20 ml of Lidocaine 2% With Epinephrine vs 40 ml 0f Lidocaine 1% With Epinephrine; Test type: Other; p = 0.48, Chi-squared

ADVERSE EVENTS:
Time Frame: 1 day
Description: The incidence of adverse effects perioperatively: nausea, dizziness, tinnitus, vomiting, convulsions or arrhythmia.
Arm/Group | 20 ml of Lidocaine 2% With Epinephrine | 40 ml 0f Lidocaine 1% With Epinephrine
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No